CLINICAL TRIAL: NCT01243905
Title: Group Psychoeducational Program for Mothers of Preschool Children With High Functional Pervasive Developmental Disorders: a Randomized Controlled Trial
Brief Title: Group Psychoeducational Program for Mothers of Children With High Functional Pervasive Developmental Disorders
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagoya City University (Other)
Responsible Party: Masako Suzuki, Nagoya City University Graduate School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCUPsychiatry003
Record Dates: First submitted 2010-11-08; First posted 2010-11-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pervasive Developmental Disorder
MeSH Terms: conditions — Child Development Disorders, Pervasive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family psychoeducation plus TAU (Active Comparator): Family psychoeducational therapy in addition to treatment as usual for the child (TAU)
  Interventions: Other: Family psychoeducational therapy plus TAU
- Treatment as usual (Placebo Comparator): Treatment as usual for the child (TAU)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Family psychoeducational therapy plus TAU — Group psychoeducation every two weeks for eight weeks in addition to treatment as usual administered by physicians
  Arms: Family psychoeducation plus TAU
Other: Treatment as usual — Treatment as usual administered by physicians
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to examine the effectiveness of group psychoeducation for the psychological distress of mothers with the children of high-functioning pervasive developmental disorder and for their behavior based on disorder traits.

DETAILED DESCRIPTION:
Pervasive Developmental Disorder (PDD) is defined by its unique symptoms such as qualitative impairment in social interaction and communication and restricted repetitive and stereotyped patterns of behavior and interests. Recently, studies have been conducted on PDD without mental retardation, and have reported that the morbidity of PDD is 0.6%-1.7％． Several studies have focused on distress of the mothers of PDD facing atypical development of their children. Some of them have indicated the associations between depression and family history of PDD. Therefore it is important to pay attention to parental mental health.

In Western countries, researchers have investigated the effectiveness of various psychotherapeutic techniques such as childcare counseling and education for mothers about how to treat their children with PDD. It has been reported that one of them which innovates pragmatical methods to manage their children and parental educational programs made improvement in parental adaptation to their children and parental mental health.

However, to the best of our knowledge, few studies have shown the effectiveness of family intervention about PDD in Japan, despite widely implementation of family psychoeducation with various approaches in medical center, public health department. New research may be needed to establish rigorous evidence base for improvement of parental mental health and of behaviors of their children with PDD.

The investigators hypothesized that psychoeducation programs for mothers in addition to treatment as usual to their children would be more effective for parental mental health and behaviors of their children with PDD than treatment usual to their children alone.

The purpose of this study is to examine the effectiveness of psychoeducation to the psychological distress of mothers with the children of high-functioning PDD and to behaviors of the children affected by disorder traits, in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers whose children have been diagnosed with any disorders by DSM-Ⅳ-TR as: 1) Autistic disorder and not mental retardation; 2) Asperger disorder; or 3) Pervasive developmental disorder not otherwise specified and not mental retardation
2. Children were diagnosed at more than 3 months before allocation
3. Children were between 2 and 6.5 years and have more than 6 months as pre-school period at allocation
4. Mothers who are native speakers of Japanese.
5. Mothers who are biological mother of and actually bringing their children.

Exclusion Criteria:

1. Mothers who are at risk of taking an emotional toll and unable to understand the contents of psychoeducation for any reason.
2. Mothers who are not allowed to participate in this study judged by the doctors of the children for any reason.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the total score of the General Health Questionaire 28(GHQ28) at 21 weeks | Baseline, 21 weeks
  GHQ:It is the shorten version of the General Health Questionaire 60. It consists four categories;somatic symptoms,anxiety and insomnia,social dysfunction and depressive tendency.

SECONDARY OUTCOMES:
Change from baseline in the total score of the General Health Questionaire 28(GHQ28) at 7 weeks | the baseline, 7weeks, 21weeks
Change from baseline in the total score of the Abnormal Behavior Checklist at 7 weeks | the baseline, 7weeks, 21weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masako Suzuki, MD, Principal Investigator — Nagoya City University Hospital
Locations (1):
- Nagoya City University Hospital, Nagoya, Aichi-ken, Japan